CLINICAL TRIAL: NCT04307576
Title: ALLTogether1 - A Treatment Study Protocol of the ALLTogether Consortium for Children and Young Adults (0-45 Years of Age) With Newly Diagnosed Acute Lymphoblastic Leukaemia (ALL)
Brief Title: A Treatment Study Protocol for Participants 0-45 Years With Acute Lymphoblastic Leukaemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mats Heyman (Other)
Collaborators: The Swedish Research Council (Other Government); The Swedish Childhood Cancer Foundation (Unknown); Pfizer (Industry); Servier (Industry); NordForsk (Unknown); Aamu Pediatric Cancer Foundation (Unknown); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other); Clinical Trial Center North (CTC North GmbH & Co. KG) (Other); Belgium Health Care Knowledge Centre (Other Government); Karolinska Institutet (Other); Cancer Research UK (Other); Fundação Rui Osório de Castro (Unknown); Acreditar - Associação de Pais e Amigos das Crianças com Cancro (Unknown); Grupo Português De Leucemias Pediátricas (Unknown); Amgen (Industry); Nova Laboratories Limited (Industry); Danish Child Cancer Foundation (Other); Danish Cancer Society (Other); The Novo Nordic Foundation (Other); Assistance Publique - Hôpitaux de Paris (Other); Direction Générale de l'Offre de Soins (Other Government); Swedish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Mats Heyman, MD, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALLTogether1
Record Dates: First submitted 2020-03-05; First posted 2020-03-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Acute Lymphoblastic
Keywords: Leukemia; Acute Leukemia; ALL; ALLTogether; Leukaemia; Inotuzumab ozogamicin; Besponsa; ALLTogether1; Blinatumomab; Blincyto; 6-tioguanine; 6-thioguanine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Imatinib Mesylate; blinatumomab

STUDY DESIGN:
Intervention Model Description: Master protocol with risk-stratification. The risk-stratified groups will proceed to non-randomised or randomised interventions in single arm (TKI) and (Blinatumomab) and parallel (R1/R2/R3) models respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- R1 - SR standard arm (No Intervention): Standard risk arm receiving standard treatment (Delayed Intensification including Doxorubicin).
- R1 - SR experimental arm (Experimental): Standard risk arm, receiving Delayed Intensification without Doxorubicin IV 3 x 30 mg/m2/dose.
  Interventions: Drug: Omitted Doxorubicin
- R2 - IR-low standard arm (No Intervention): Standard treatment with Delayed Intensification including Doxorubicin and Maintenance including Vincristine+Dexamethasone pulses.
- R2 - IR-low experimental arm A (Experimental): Standard treatment with omission of Doxorubicin IV 3 x 30 mg/m2/dose in the Delayed Intensification phase.
  Interventions: Drug: Omitted Doxorubicin
- R3 - IR-high standard arm (No Intervention): Intermediate risk high arm receiving Standard Maintenance Therapy.
- R3-InO - IR-high experimental arm (Experimental): Inotuzumab IV 0,5 mg/m2, given on days 253, 260, 267 and on days 274, 281, 288 before start of Standard Maintenance Therapy.
  Interventions: Drug: Inotuzumab Ozogamicin+Standard Maintenance Therapy
- ABL-class fusions intervention (Experimental): Imatinib p.o. 340 mg/m2 given daily from day 15 or 30 (depending on age) to the end of therapy (week 106) in addition to Standard IR-high chemotherapy.
  Interventions: Drug: Imatinib
- R3-TEAM - IR-high experimental arm (Experimental): 6-tioguanine p.o, 2,5-12,5 mg/m2, given daily in addition to Standard Maintenance Therapy.
  Interventions: Drug: 6-tioguanine+Standard Maintenance Therapy
- ALLTogether1 DS Blinatumomab intervention (Experimental): Blinatumomab IV, 5 mcg/m2/day up to 28 mcg/day (detailed dosing in protocol) continous infusion. Two 28 day courses with a two week treatment free interval in between. Blinatumomab courses replace Consolidation 1 and Consolidation 2 in the standard protocol adapted for Down syndrome patients.
  Interventions: Drug: Blinatumomab
- R2 - IR-low experimental arm B (Experimental): Standard treatment with omission of monthly pulses of Vincristine IV 1,5 mg/m2/dose and 5 days of Dexamethasone p.o. 6 mg/m2/day in the Maintenance Phase.
  Interventions: Drug: Omitted Vincristine+Dexamethasone pulses

INTERVENTIONS:
Drug: Omitted Doxorubicin — Omission of IV Doxorubicin
  Arms: R1 - SR experimental arm; R2 - IR-low experimental arm A
Drug: Omitted Vincristine+Dexamethasone pulses — Omission of Vincristine+Dexamethasone pulses
  Arms: R2 - IR-low experimental arm B
Drug: Inotuzumab Ozogamicin+Standard Maintenance Therapy — Addition of IV Inotuzumab ozogamicin before Maintenance Therapy
  Other Names: Besponsa+Maintenance Therapy
  Arms: R3-InO - IR-high experimental arm
Drug: Imatinib — p.o. Imatinib
  Arms: ABL-class fusions intervention
Drug: 6-tioguanine+Standard Maintenance Therapy — Addition of p.o. 6-tioguanine to Standard Maintenance Therapy
  Arms: R3-TEAM - IR-high experimental arm
Drug: Blinatumomab — IV Blinatumomab
  Other Names: Blincyto
  Arms: ALLTogether1 DS Blinatumomab intervention

SUMMARY:
ALLTogether collects the experience of previously successful treatment of infants, children and young adults, with ALL from a number of well-renowned study groups into a new master protocol, which is both a comprehensive system for stratification and treatment of ALL in this age-group as well as the basis for several randomised and interventional trials included in the study-design.

DETAILED DESCRIPTION:
ALLTogether is a European clinical treatment study for acute lymphoblastic leukaemia (ALL) in infants, children and young adults. The aims are to improve survival and quality of survival. In young people, ALL has excellent outcome with an overall survival of about 92% in children and 75% in young adults. Infants with BCP-ALL and KMT2A-rearrangements have a worse outcome and are treated according to separate protocols, but infants with KMT2A-germline and T-cell ALL have acceptable outcome on standard ALL therapy. However, patients still die of disease - from relapse because of under-treatment and a large fraction of patients are also over-treated: All patients risk treatment-related death and some suffer long-term side-effects or secondary cancer. To show improvement with such good survival, large populations are needed.

Study groups from Sweden, Norway, Iceland, Denmark, Finland, Estonia and Lithuania (NOPHO), the UK (UKALL), the Netherlands (DCOG), Germany (COALL), Belgium (BSPHO), Portugal (SHOP), Ireland (PHOAI), and France (SFCE), have designed a common treatment protocol.

The study has a complex clinical trial design with sub-protocols (the randomisations / intervention) connected to a master protocol. The master protocol consists of well established therapy-elements and in its design typical for current ALL therapy. The master protocol therapy is in the study design considered as standard of care (SOC) therapy for infants, children and young adults with ALL.

The study structure is defined by a master protocol onto which randomised and interventional sub-protocols as well as sub-studies may be added, run and stop in a modular fashion.

The randomisations / intervention may identify therapy that is less toxic, but equally efficacious for sub-groups of patients and innovative therapy that may reduce relapses and death from ALL. In the master protocol, improved risk-stratification is likely to increase survival and reduce unnecessary toxicity and the introduction of therapeutic drug monitoring (TDM) of Asparaginase activity will make the use of Asparaginase more rational and efficient and may thus improve overall outcomes.

The investigators hypothesise that patients stratified to the standard-risk group are over-treated. Therefore, it will be tested if the treatment can be safely reduced. In the R1 randomisation, patients will be randomised to receiving the Delayed Intensification (DI) phase of therapy with or without the anthracycline Doxorubicin.

A similar hypothesis of over-treatment will also be tested in patients stratified to the intermediate risk-low group. In the R2 randomisation patients will be randomly assigned to either removal of Doxorubicin during the DI phase or removal of Vincristine and Dexamethasone pulses during the maintenance phase or to the control group, which will be treated with Doxorubicin in DI as well as Vincristine and Dexamethasone pulses during maintenance. Patients will only be randomised once.

Randomisation R1 and R2 are only considered for children since adults have worse outcome and very poor survival after relapse, but the risk-stratification is likely to reduce the number of high-risk cases also in the adult-group.

Patients stratified as intermediate risk-high (IR-high) are identified as having an increased risk of relapse and thus a less favourable prognosis than the standard- and intermediate risk-low groups, but a more favourable prognosis than the high risk patients. The majority of all relapses in childhood ALL is expected to occur in the IR-high group. Following a relapse, only approximately 40% of the children can be successfully treated again and for adults the corresponding figure is less than 20 %, so preventing relapses is very important. New treatment options that improves the antileukaemic efficacy and which have an improved safety profile are urgently needed.

For IR-high patients Randomisation 3 (R3) is available. In R3 patients will be randomised to receive either:

1. the first six weeks of maintenance treatment are replaced by two 3- week cycles of Inotuzumab ozogamicin (InO) - Besponsa®. This is followed by maintenance therapy similar to the standard arm.
2. the addition of low dose 6-tioguanine (6TG) as an addition to the standard maintenance therapy.
3. standard maintenance therapy.

Patients with ABL-class fusions in their leukaemic clone will, as a non-randomised experimental intervention, be treated with an addition of a tyrosine-kinase inhibitor during the induction phase (for patients <25 years) and from the consolidation phase (patients ≥25 years). This intervention may shift therapy for previously resistant cases to lower intensity treatment with the associated reduced morbidity and may also reduce the number of relapses in analogy with the results in Ph+ ALL. The reason for not performing a randomised comparison is the rarity of the aberration and also the diversity of ABL-class fusions, reducing statistical power for any comparison further. For this reason, the results of this intervention may be pooled with other study-groups trying similar approaches.

A new intervention is introduced for Down syndrome patients with CD19 positive ALL: ALLTogether1 DS (NRI2). For Down syndrome-ALL patients who have end of Induction MRD detectable but <25% two conventional chemotherapy consolidation blocks will be replaced with two blocks of Blinatumomab. Recruitment to this intervention was closed at the end of August 2024.

For high-risk B-lineage patients, CAR-T therapy can be an alternative to high-risk blocks and stem-cell transplant, but in this case the intervention (CAR-T infusion) will be performed outside the ALLTogether1 study. However, the stratification-system in ALLTogether1 will define the population with a potential CAR-T indication.

ALLTogether1 also includes five sub-studies:

Efficacy and pharmacokinetics of Imatinib in ABL-class fusion positive ALL

Target population: All ABL-class patients enrolled in the ALLTogether study. Biomaterials to be collected at diagnosis, during TKI treatment, follow-up and relapse.

Aims

1. To determine the efficacy and dosing target of imatinib in the treatment of ABL-class leukemia
2. To find the best discriminative biomarkers for TKI response in ABL-class ALL
3. To determine the frequency of intrinsic (at diagnosis) and acquired TKI resistance (due to treatment), including backtracking of mutations using imatinib PK/PD findings during treatment
4. To find causes of TKI resistance in ABL-class patients
5. To describe the pharmacokinetics of Imatinib in TKI-treated patients

Objectives

1. To determine the percent of ABL-class patients who need to switch from IR-high to HR because of high MRD levels
2. To determine the effect of imatinib exposure on clinical outcome, including pharmacokinetic measurements of imatinib
3. To determine the molecular response to imatinib by monitoring fusion gene levels and mutational spectrum at diagnosis and during follow up
4. To determine whether the molecular response parameters reflect the Ig/TCR MRD or flow-MRD response or are a better predictor of therapy failure than Ig/TCR or flow-based MRD monitoring
5. To determine the phosphorylation status of ABL-class proteins and presence of TKI-resistance associated mutations in ABL genes prior to imatinib treatment and the emergence of such mutations during treatment with imatinib
6. To determine the presence of mutations in regulatory /other genes before and during imatinib treatment and functionally address the importance of these mutations in TKI resistance
7. To determine whether the efficacy of TKIs depends on the type of fusion gene
8. To describe inter- and intraindividual variations in imatinib PK (=trough levels) during therapy of ABL-class ALL
9. To describe associations between PK of imatinib and end-of-induction MRD (<25 yrs only) and end-of-consolidation MRD (all patients)
10. To describe associations between imatinib PK and relapse rates (overall, bone-marrow and CNS), event-free survival as well as overall survival;
11. To describe associations between imatinib PK and toxicities (including e.g. height z-scores at diagnosis and end of therapy, pancreatitis, treatment delays) with focus on those toxicities that are routinely monitored in ALLTogether.

Biomarkers to Reform Approaches to therapy-Induced Neurotoxicity (BRAIN)

Target population: All patients registered on ALLTogether1 aged ≥ 4 years at end of therapy (Arm A) and all patients registered on ALLTogether1 aged 2-21 years at start of therapy (Arm B) and without:

1. Pre-existing neurodevelopmental delay (e.g Trisomy 21) prior to diagnosis of ALL
2. Significant visual or motor impairment preventing use of a computer/touch screen ipad

All centres are invited to enrol to arm A (Main BRAIN) of the study. Arm B (Longitudinal BRAIN) will be carried out in selected centres.

Aims

1. To implement universal screening of all children for adverse neurocognitive outcomes at the end of treatment using a validated user-friendly computer software programme (CogState) and compare neurocognitive outcomes by treatment allocation (Arm A).
2. To identify risk factors for adverse outcomes including whether acute neurotoxic events are associated with poor performance on cognitive tests at end of therapy compared to patients without acute neurotoxicity (Arm A).
3. To examine changes in neurocognitive performance over time and the risk/protective factors associated with differences in outcome, such as demographic, clinical, and physical/psychosocial factors (Arm B).

Primary end-point

a. Proportion of children with a z-score <1.5 on detection and/or identification CogState tasks in each treatment arm at the end of ALL therapy. A z-score < 1.5 correlates with moderate cognitive impairment at a level that may require additional support.

Secondary and exploratory end-points

1. Association between CogState scores at end of treatment and overt neurotoxic episodes as recorded on the trial adverse event database.
2. Association between Cogstate scores and clinical and demographic variables - age, sex, ethnicity, CNS status.
3. Proportion of children with scores <1.5SD for one card learning (learning), one back (working memory), Groton's maze (executive function), digit symbol substitution (processing speed) on different treatment arms.
4. Association between CogState scores and patient reported outcome measures/Quality of life measurements collected as part of the main ALLTogether1 trial.
5. Changes in neurocognitive scores over time, including CogState and BRIEF-2/BRIEF-A scores.
6. Association between neurocognitive scores over time and interactions with demographic variables (age, sex), clinical variables (treatment arm, neurotoxicity), social-emotional and physical functioning (SDQ, PedsQL 4.0 Generic; PedsQL 3.0 Fatigue), and family factors (MEES; PedsQL FIM).

Association between asparaginase activity levels and outcome

Target population: All patients included in the ALLTogether1 protocol are eligible for participation.

Primary aim

To study the association between asparaginase activity levels and outcome (MRD, relapse, survival)

Secondary aims

1. To evaluate the association between asparaginase activity levels and toxicities, such as pancreatitis, infections and deep venous thrombosis (DVT)
2. To evaluate the association between asparaginase activity levels and hepatotoxicity in a subset of patients

CSF-Flow

Target population: All patients included in the ALLTogether1 protocol are eligible for participation

Aims

1. To use cerebrospinal fluid (CSF) flow cytometry (FCM) to improve the accuracy of diagnostic tests for CNS leukaemia compared to conventional CSF cytology. An associated objective will be to develop a recommended protocol for CSF flow cytometry with external quality assessment to ensure uniformity of measurement across the ALLTogether consortium.
2. To investigate whether negative FCM identifies a group of children at very low risk of CNS relapse, suitable for testing de-escalation of CNS-directed therapy in future trials.
3. To investigate whether positive FCM can identify children at increased risk of CNS relapse and whether patients with persistent positivity (FCM positive at day 15 onwards) might benefit from studies testing escalated CNS-directed therapy or a switch to more intensive treatment arms.
4. To collect matching CSF supernatant for studies comparing CSF FCM with soluble biomarkers (e.g. metabolic, cell-free DNA, proteomic and microRNA).

Maintenance therapy pharmacokinetics/-dynamics study

Target population: All patients included in the ALLTogether1 protocol are eligible for participation. For IR-high patients participating in the randomised InO- and TEAM sub-protocols, the monitoring of 6-mercaptopurine (6MP)/Methotrexate (MTX) metabolites at three months intervals is mandatory.

Aims and specific objectives

1. To map pharmacokinetics of 6MP and MTX during maintenance therapy in all patients in the ALLTogether protocol.
2. To associate metabolite profiles with TPMT and NUDT15 variants, as routinely analysed in ALLTogether.
3. To explore the association of event-free survival with DNA-TG and other 6MP/MTX metabolites.
4. To explore the association between risk of second cancers with DNA-TG and other 6MP/MTX metabolites.
5. To explore the association of risk of invasive infections with DNA-TG and other 6MP/MTX metabolites.
6. To explore the association of risk of osteonecrosis with DNA-TG and other 6MP/MTX metabolites.
7. To explore the association of sinusoidal obstruction syndrome with DNA-TG and other 6MP/MTX metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed with T-lymphoblastic (T-cell) or B-lymphoblastic precursor (BCP) leukaemia (ALL) according to the WHO-classification of Tumours of Haematopoetic and Lymphoid Tissues (Revised 4th edition 2017) and with a diagnosis confirmed by an accredited laboratory at a participating paediatric oncology or adult haematology centre.
* Age 0 - < 46 years (one day before 46th birthday) at the time of diagnosis with the exception of infants with KMT2A-rearranged (KMT2A-r) BCP ALL.
* Patients with surface immunoglobulin negative (sIG-) BCP-ALL and an IG::MYC rearrangement, unless they have a concurrent BCL2/6 rearrangement. T-ALL patients with MYC translocations.
* Informed consent signed by the patient and/or parents/legal guardians according to country-specific age-related guidelines.
* The ALL diagnosis should be confirmed by an accredited laboratory at a participating paediatric oncology or adult haematology centre.
* The patient should be diagnosed and treated at a participating paediatric oncology or adult haematology centre in the participating countries.
* The patient should be a resident in one of the participating countries on a permanent basis or should intend to settle in a participating country, for instance by an application for asylum. Patients who are visiting the country as tourists should not be included. However, returning expatriots with primary diagnosis abroad may be included if no treatment has been administered and the diagnostic procedures are repeated at a participating centre.
* All women of childbearing potential (WOCBP) have to have a negative pregnancy test within 2 weeks prior to the start of treatment.
* For each intervention/randomisation an additional set of inclusion-criteria is provided.

Exclusion Criteria:

* Age < 365 days and KMT2A-rearranged (KMT2A-r) BCP-ALL (documented presence of a KMT2A-split by FISH and/or a KMT2A fusion transcript).
* Age >45 years at diagnosis.
* Patients with a previous malignant diagnosis (ALL as a second malignant neoplasm - SMN).
* Relapse of ALL.
* Patients with mature B-ALL (as defined by surface IG positivity) or any patients with IG::MYC and a concurrent BCL2/6 rearrangement.
* Patients with Ph-positive ALL (documented presence of t(9;22)(q34;q11) and/or of the BCR::ABL fusion transcript). These patients will be transferred to an appropriate trial for t(9;22) if available.
* Previously known ALL prone syndromes (e.g. Li-Fraumeni syndrome, germline ETV6 mutation), except for Down syndrome. Exploration for such ALL prone syndromes is not mandatory and patients in whom genetic work-up reveals a new germ-line mutation (index-cases) will remain in the study.
* Treatment with systemic corticosteroids corresponding to (>10mg prednisolone/m2/day) for more than one week and/or other chemotherapeutic agents in a 4-week interval prior to diagnosis (pre-treatment).
* Pre-existing contraindications to any treatment according to the ALLTogether protocol (constitutional or acquired disease prior to the diagnosis of ALL preventing adequate treatment).
* Any other disease or condition, as determined by the investigator, which could interfere with the participation in the study according to the study protocol, or with the ability of the patients to cooperate and comply with the study procedures.
* Women of childbearing potential who are pregnant at the time of diagnosis.
* Women of childbearing potential and fertile men who are sexually active and are unwilling to use adequate contraception during therapy. Efficient birth control is required.
* Female patients, who are breast-feeding.
* Essential data missing from the registration of characteristics at diagnosis (in consultation with the protocol chair).
* For each intervention/randomisation an additional set of exclusion-criteria is provided.

Ages: 0 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6430 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) for the whole protocol | 5 year estimates from the time of diagnosis will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  The primary endpoint for the whole protocol (compared with the legacy protocols of the participating study-groups forming the consortium) is event-free survival (EFS) - as defined in the protocol.
Event-free survival (EFS) for the TKI intervention | From the start of TKI (day 15 or day 30), 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up for all interventions except Inotuzumab-randomisation (minimum 2-year follow-up).
  The primary endpoint for the TKI intervention is event-free survival (EFS) - as defined in the protocol, from the start of TKI until event or end of follow-up
Disease-free survival (DFS) R1 + R2 | 5 and 8 year estimates from the time of randomisation will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  The primary endpoint for Randomisation 1 and 2 is disease-free survival (DFS) - as defined in the protocol counting from the time of randomisation
Disease-free survival (DFS) R3 | 5 year estimates from the time of randomisation will be measured but adequate follow-up for these estimates will be ensured: at least 2-year follow-up
  The primary endpoint for Randomisation 3 and the ABL-class fusion intervention is disease-free survival (DFS) - as defined in the protocol counting from the time of randomisation (R3) and the start of TKI-therapy (ABL-class fusion intervention).
MRD response after 1 cycle of Blinatumomab | End of first Blinatumomab infusion +/- 1 week
  Fraction of patients with undetectable MRD ("Complete MRD response") at the end of one cycle of Blinatumomab (+/- 1 week)

SECONDARY OUTCOMES:
Overall survival (OS) for the whole protocol | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Overall survival defined as time from diagnosis to death or end of follow-up for surviving patients.
Overall survival (OS) for R1 + R2 | 5 and 8 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Overall survival defined as time from randomisation to death or end of follow-up for surviving patients.
Overall survival (OS) for R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Overall survival defined as time from randomisation to death or end of follow-up for surviving patients.
Overall survival (OS) for R3-TEAM associated with DNA-TG | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Overall survival as defined above in relation to DNA-TG.
Overall survival (OS) for TKI | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up (TKI).
  Overall survival defined as time from start of TKI to death or end of follow-up for surviving patients
Overall survival (OS) for ALLTogether1 DS | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Overall survival defined as time from start of Blinatumomab to death or end of follow-up for surviving patients
Induction death | From diagnosis until death before remission (at the earliest, day 29) or in case of no CR day 29, completion of induction and consolidation 1 (protocol day 99 - Down) and in addition 3 high-risk blocks (protocol day 134 - all other patients)
  Fraction of patients who die as well as cumulative incidence of death before achieved complete remission (CR) within the time-frame described in the protocol
Resistant disease | From diagnosis until achieved complete remission (at the earliest, day 29) or in case of no CR day 29, assessment after induction and consolidation 1 (protocol day 99-Down patients) and in addition 3 high-risk blocks (protocol day 134-all other patients)
  Fraction of patients as well as cumulative incidence of resistant disease as described in the protocol. Induction death as competing risk.
Cumulative incidence of relapse for the whole protocol | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from achieved complete remission until relapse as defined in the protocol or end of follow-up. Second malignancy, death in complete remission as competing events.
Cumulative incidence of relapse for R1 + R2 | 5 and 8 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from randomisation until relapse as defined in the protocol or end of follow-up. Second malignancy, death in complete remission as competing events.
Cumulative incidence relapse for R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Time from randomisation until relapse as defined in the protocol or end of follow-up. Second malignancy, death in complete remission as competing events.
Cumulative incidence relapse for R3-TEAM in association with DNA-TG | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Cumulative incidence of relapse as defined for R3 in association with DNA-TG for R3-TEAM. Second malignancy, death in complete remission as competing events.
Cumulative incidence CD22 negative relapse for R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Time from randomisation until relapse without expression of CD22 as defined in the protocol or end of follow-up. Second malignancy, death in complete remission and relapse with CD22 expression as competing events.
Cumulative incidence relapse for TKI | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of TKI until relapse as defined in the protocol or end of follow-up. Second malignancy, death in complete remission as competing events.
Cumulative incidence relapse for ALLTogether1 DS | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of Blinatumomab until relapse as defined in the protocol or end of follow-up. Second malignancy, death in complete remission as competing events.
Cumulative incidence of CD19 negative relapse for ALLTogether1 DS | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of Blinatumomab until CD19 negative relapse as defined in the protocol or end of follow-up. Second malignancy, death in complete remission and CD19 positive relapse as competing events.
Cumulative incidence of second malignant neoplasm (SMN) for the whole protocol | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from achieved complete remission until diagnosis of second malignant neoplasm as defined in the protocol or end of follow-up. Relapse and death in complete remission as competing events.
Cumulative incidence of second malignancy for R1+R2 | 5 and 8 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from randomisation until diagnosis of second malignant neoplasm as defined in the protocol or end of follow-up. Relapse and death in complete remission as competing events.
Cumulative incidence of second malignancy for R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up.
  Time from randomisation until diagnosis of second malignant neoplasm as defined in the protocol or end of follow-up. Relapse and death in complete remission as competing events.
Cumulative incidence of second malignancy for R3-TEAM in association with DNA-TG | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up.
  Cumulative incidence of second malignancy as defined above for R3 in association with DNA-TG for R3-TEAM. Relapse and death in complete remission as competing events.
Cumulative incidence of second malignancy for TKI | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from start of TKI until diagnosis of second malignant neoplasm as defined in the protocol or end of follow-up. Relapse and death in complete remission as competing events.
Cumulative incidence of second malignancy for ALLTogether1 DS | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from start of Blinatumomab until diagnosis of second malignant neoplasm as defined in the protocol or end of follow-up. Relapse and death in complete remission as competing events.
Cumulative incidence of death in complete remission for the whole protocol | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from achieved complete remission until death in complete remission as defined in the protocol or end of follow-up. Relapse and second malignant neoplasm as competing events.
Cumulative incidence of death in complete remission for R1+R2 | 5 and 8 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up.
  Time from randomisation until death in complete remission as defined in the protocol or end of follow-up. Relapse and second malignant neoplasm as competing events.
Cumulative incidence of death in complete remission for R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Time from randomisation until death in complete remission as defined in the protocol or end of follow-up. Relapse and second malignant neoplasm as competing events.
Cumulative incidence of death in complete remission for TKI | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of TKI until death in complete remission as defined in the protocol or end of follow-up. Relapse and second malignant neoplasm as competing events.
Cumulative incidence of death in complete remission for ALLTogether1 DS | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of Blinatumomab until death in complete remission as defined in the protocol or end of follow-up. Relapse and second malignant neoplasm as competing events.
Cumulative incidence of treatment-related mortality for the whole protocol | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from diagnosis until death during induction, death in complete remission or death from second malignant neoplasm (if not related to SMN-treatment).
Cumulative incidence of treatment-related mortality R1+R2 | 5 and 8 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up.
  Time from randomisation until death in complete remission or death from second malignant neoplasm (if not related to SMN-treatment).
Cumulative incidence of treatment-related mortality R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Time from randomisation until death in complete remission or death from second malignant neoplasm (if not related to SMN-treatment).
Cumulative incidence of treatment-related mortality TKI | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of TKI until death in complete remission or death from second malignant neoplasm (if not related to SMN-treatment).
Leukaemia specific mortality for the whole protocol | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from diagnosis until death after resistant disease or relapse - as defined in the protocol.
Leukaemia specific mortality for R1+R2 | 5 and 8 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up.
  Time from randomisation until death after relapse - as defined in the protocol.
Leukaemia specific mortality for R3 | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 2 years follow-up
  Time from randomisation until death after relapse - as defined in the protocol.
Leukaemia specific mortality for TKI | 5 year estimates will be measured but adequate follow-up for these estimates will be ensured: at least 5 years follow-up
  Time from start of TKI until death after relapse - as defined in the protocol.
Incidence of Adverse Events of Special Interest (AESIs) per treatment-phase in the whole protocol and TKI intervention | From time of diagnosis after each treatment-phase (one extra in the middle of maintenance) and annually until 5 years from discontinuation of therapy.
  Cumulative incidence of 19 AESIs as defined in the protocol
Incidence of Adverse Events of Special Interest (AESIs) extra assessment (R1+R2) | Cumulative incidence of AESIs estimated 3 months after start of maintenance (R1+R2) and at the end of maintenance (R2)
  Cumulative incidence of 4 additional AESIs as defined in the protocol
Incidence of Adverse Events of Special Interest (AESIs) extra assessment (R3) | Cumulative incidence of AESIs estimated at the end of maintenance.
  Cumulative incidence of 3 additional AESIs as defined in the protocol
Incidence of Serious Adverse Events (SAEs) and Adverse Events (AEs) related to R3 | From time of randomisation until the end of maintenance therapy (approximately 77 weeks from randomisation)
  Cumulative incidence of SAEs and AEs (with limitations) as defined in the protocol
Quantitative measures of toxicity R1+R2 | From time of randomisation, assessment after delayed intensification and 6 weeks after start of maintenance
  Days: in hospital, with iv antibiotics, with iv analgesics, with iv nutritional support
Metabolic consequences of steroid exposure (R2) | At the end of therapy (approximately 94 weeks from randomisation) and 5 years after discontinuation of treatment
  Measurements of BMI
Association of Disease-free survival (DFS) with DNA-TG for R3-TEAM | 5 year estimates from the time of randomisation will be measured but adequate follow-up for these estimates will be ensured: at least 2-year follow-up
  Disease-free survival (DFS) - as defined above associated with DNA-TG.
Cumulative incidence of Sinusoidal Obstruction Syndrome (SOS) and Nodular Regenerative Hyperplasia (NRH) for R3-TEAM | Cumulative incidence of SOS/NRH estimated at the end of follow-up.
  Time from randomisation until diagnosis of SOS or NRH as defined in the protocol or end of follow-up.
Cumulative incidence of Osteonecrosis for R3-TEAM | Cumulative incidence of osteonecrosis estimated at the end of follow-up.
  Time from randomisation until diagnosis of osteonecrosis as defined in the protocol or end of follow-up.
Event-free survival (EFS) for ALLTogether1 DS | From the start of Blinatumomab, 5 year estimate will be measured but adequate follow-up for this estimate will be ensured: at least 5 years follow-up.
  Event-free survival as defined in the protocol, from the start of Blinatumomab until death from any cause, relapse, second malignancy, protocol therapy failure (MRD>1% after 2 cycles blinatumomab and Augmented BFM consolidation) or end of follow-up.
Incidence of Blinatumomab refractory disease for ALLTogether1 DS | From the start of Blinatumomab until end of 2nd cycle of Blinatumomab (each cycle is 4 weeks followed by a 2-week treatment free period)
  Incidence of progressive disease under Blinatumomab treatment or MRD ≥1% at the end of the 2nd cycle of Blinatumomab.
Incidence of Protocol Therapy Failure for ALLTogether1 DS | From the start of Blinatumomab until the end of Consolidation 1 (85-140 days: 15-70 days of Blinatumomab therapy + 70 days of Consolidation 1)
  Incidence of patients who have MRD ≥1 % post 2 cycles of Blinatumomab followed by Augmented BFM consolidation, corresponding to original protocol day 99, or unchanged/increasing MRD during Augmented BFM consolidation corresponding to original protocol day 57.

OTHER OUTCOMES:
6-mercaptopurine and Methotrexate metabolite pharmacokinetics (i.e. Ery-TGN/MeMP/MTXpg) for R3-TEAM | From start of Maintenance therapy until the end of Maintenance therapy (protocol week 38 until protocol week 108)
  Measurements of metabolites Ery-TGN/MeMP/MTXpg during Maintenance therapy.
Abnormal liver function parameters (including hypoglycemia) for R3-TEAM | From start of Maintenance therapy until the end of Maintenance therapy (protocol week 38 until protocol week 108)
  Liver function parameters including hypoglycemia during Maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mats Heyman, MD, PhD, Study Chair — Karolinska University Hospital
Locations (130):
- Belgium (7):
  - L'hôpital Universitaire des enfants Reine Fabiola (Huderf), Brussels
  - Cliniques Universitaires Saint-Luc (UCL), Brussels
  - University Hospital Antwerp, Edegem
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Dept of Paediatrics, Leuven
  - CHC MontLégia, Boulevard Patience et Beaujonc 2, Liège
  - CHR de la Citadelle, Liège
- Denmark (6):
  - Aalborg University Hospital, Dept of Paediatrics, Aalborg
  - Aarhus University Hospital, Aarhus
  - Aarhus University Hospital, Child and Adolescent Health, Aarhus
  - Rigshospitalet, Dept of Haematology, Copenhagen
  - Rigshospitalet, Dept of Paediatrics, Copenhagen
  - Odense University Hospital, Dept of Paediatrics, Odense
- Estonia (3):
  - North Estonia Medical Centre, Dept of Haematology, Tallinn
  - Tallinn Children´s Hospital, Dept of Paediatrics, Tallinn
  - Tartu University Hospital, Tartu
- Finland (10):
  - Helsinki University Hospital, Dept of Haematology, Helsinki
  - Helsinki University Hospital, Dept of Paediatrics, Helsinki
  - Kuopio University Hospital, Dept of Haematology, Kuopio
  - Kuopio University Hospital, Dept of Paediatrics, Kuopio
  - Oulu University Hospital, Dept of Haematology, Dept of Medicine, Oulu
  - Oulu University Hospital, Dept of Paediatrics, Oulu
  - Tampere University Hospital, Dept of Haematology, Tampere
  - Tampere University Hospital, Dept of Paediatrics, Tampere
  - Turku University Hospital, Clinical Haematology and Stem Cell Transplantation Unit, Turku
  - Turku University Hospital, Dept of Paediatrics, Turku
- France (29):
  - CHU Amiens Groupe Hospitalier Sud, Amiens
  - CHU Angers, Angers
  - CHRU Besançon, Besançon
  - CHU Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - CHRU Brest - Morvan, Brest
  - Centre Hospitalier Universitaire Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon Hôpital François Mitterrand, Dijon
  - CHU de Grenoble site Nord - Hôpital Albert Michallon, Grenoble
  - CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la mère et de l'enfant, Limoges
  - CHU de Lyon HCL - GH Est-Institut d'hématologie et d'oncologie pédiatrique IHOP, Lyon
  - CHU de Marseille - Hôpital de la Timone, Marseille
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes-Hôpital enfant-adolescent, Nantes
  - CHU Nice - Hôpital l'Archet 2, Nice
  - CHU Paris Saint Louis, Paris
  - CHU Paris Armand Trousseau, Paris
  - CHU Paris - Hôpital Robert Debré, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims-American Hospital, Reims
  - CHU Rennes - Hôpital sud, Rennes
  - CHU Rouen, Rouen
  - CHU De La Réunion - Site Nord (Hôpital Félix GUYON), Saint-Denis
  - CHU Saint Etienne Hôpital Nord, Saint-Etienne
  - CHU Strasbourg -Hôpital de Hautepierre, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Tours- Hôpital Clocheville, Tours
  - CHU de Nancy - Hôpital de Brabois Enfant, Vandœuvre-lès-Nancy
- Germany (6):
  - Evangelisches Klinikum Bethel, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Bremen Mitte, Bremen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - HELIOS Klinikum Krefeld, Krefeld
  - Universitätsmedizin Mainz, Mainz
- Landspitali University Hospital, Children's Hospital, Reykjavik, Iceland
- Our Lady's Children's Hospital, Dublin, Ireland
- Lithuania (2):
  - Children's Hospital, Affiliate of Vilnius University Hospital Santaros Klinikos, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Netherlands (2):
  - Princess Máxima Center for Pediatric Oncology, Utrecht
  - University Medical Center Utrecht, Utrecht
- Norway (9):
  - Haukeland University Hospital, Dept of Haematology, Bergen
  - Haukeland University Hospital, Dept of Paediatrics, Bergen
  - Oslo University Hospital, Dept of Haematology, Oslo
  - Oslo University Hospital, Dept of paediatric haemato- and oncology, Oslo
  - Stavanger University Hospital, Dept of Haematology, Stavanger
  - University Hospital North Norway, Dept of Haematology, Tromsø
  - University Hospital of North Norway, Dept of Paediatrics, Tromsø
  - St. Olavs University Hospital, Dept of Paediatrics, Trondheim
  - St. Olavs University Hospital, Dept of Haematology, Trondheim
- Portugal (3):
  - Centro Hospitalar e Universitário de Coimbra, EPE - Hospital Pediátrico de Coimbra, Coimbra
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Sweden (13):
  - Sahlgrenska University Hospital, Section for Haematology and coagulation, Gothenburg
  - Sahlgrenska University Hospital, Dept of Paediatric Haematology and Oncology, Gothenburg
  - Linköping University Hospital, Dept of Haematology, Linköping
  - Linköping University Hospital, Dept of Paediatrics, Linköping
  - Skåne University Hospital, Dept of Haematology, Lund
  - Skåne University Hospital, Dept of Paediatrics, Lund
  - Örebro University Hospital, Section for Haematology, Örebro
  - Karolinska University Hospital, Dept of Paediatric Oncology and Haematology, Stockholm
  - Karolinska University Hospital, Patient area Haematology, Stockholm
  - Norrland University Hospital, Dept of Haematology, Umeå
  - Norrland University Hospital, Dept of Paediatrics, Umeå
  - Uppsala University Hospital, Dept of Haematology, Uppsala
  - Uppsala University Hospital, Dept of Paediatric Haematology and Oncology, Uppsala
- United Kingdom (38):
  - Aberdeen Royal Infirmary, Aberdeen, Aberdeen
  - Royal Aberdeen Children's Hospital, Aberdeen, Aberdeen
  - Royal Belfast Hospital for Sick Children, Belfast, Belfast
  - Belfast City Hospital, Belfast, Belfast
  - The Queen Elizabeth Hospital, Birmingham, Birmingham
  - Birmingham Children's Hospital, Birmingham, Birmingham
  - Bristol Royal Hospital for Children / Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge, Cambridge
  - Noah's Ark Children's Hospital for Wales, Cardiff, Cardiff
  - University Hospital of Wales, Cardiff, Cardiff
  - Ninewells Hospital, Dundee, Dundee
  - Western General Hospital, Edinburgh, Edinburgh
  - Royal Hospital for Children and Young People, Edinburgh, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow, Glasgow
  - Royal Hospital for Children, Glasgow, Glasgow
  - Leeds General Infirmary, Leeds, Leeds
  - Leeds St James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester, Leicester
  - Alder Hey Children's Hospital, Liverpool, Liverpool
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - University College London Hospital, London, London
  - Great Ormond Street Hospital for Children, London, London
  - King's College Hospital, London
  - St. Bartholomews Hospital, London
  - Royal Manchester Children's Hospital, Manchester, Manchester
  - The Christie NHS Foundation Trust (PTC), Manchester
  - Freeman Hospital, Newcastle, Newcastle
  - Royal Victoria Infirmary, Newcastle, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Nottingham Queen's Medical Centre, Nottingham
  - Churchill Hospital, Oxford, Oxford
  - John Radcliffe Hospital, Oxford, Oxford
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield, Sheffield
  - Sheffield Children's Hospital, Sheffield, Sheffield
  - Southampton General Hospital, Southampton, Southampton
  - Royal Stoke University Hospital, Stoke, Stoke
  - Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
ALLTogether Data Sharing Policy FINAL VERSION 1.0 DATED 12APRIL2022 applies (full details available from Trial Central Office):
  Policy
  1. The ALLTogether Consortium aims to maximise the availability of research data to the academic community for academic non-commercial research purposes with as few restrictions as possible.
  2. All research papers should be open access whenever possible.
  3. Clinical data: The ALLTogether Consortium will consider requests for individual participant data (IPD) that underlie published results after deidentification. Requests for access for unpublished data will also be considered on a case-by-case basis.
  4. ALLTogether scientific data underpinning basic science/translational research papers should be made available to other researchers in the ALLTogether consortium and requests from academic researchers outside the consortium for access to scientific datasets should be addressed to the lead investigator of the ALLTogether study.
Supporting Information: Study Protocol, SAP
Time Frame: The ALLTogether Consortium will consider requests for individual participant data (IPD) that underlie published results after deidentification. Requests for access for unpublished data will also be considered on a case-by-case basis.
Access Criteria: Data access requests will be reviewed by The ALLTogether Board and, when applicable the ALLTogether Scientific committee.
  IPD will only be released if all personalised identifiers can be removed and for the sole use of the approved request (tertiary dissemination will not be permitted).
  Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Toft N, Birgens H, Abrahamsson J, Griskevicius L, Hallbook H, Heyman M, Klausen TW, Jonsson OG, Palk K, Pruunsild K, Quist-Paulsen P, Vaitkeviciene G, Vettenranta K, Asberg A, Frandsen TL, Marquart HV, Madsen HO, Noren-Nystrom U, Schmiegelow K. Results of NOPHO ALL2008 treatment for patients aged 1-45 years with acute lymphoblastic leukemia. Leukemia. 2018 Mar;32(3):606-615. doi: 10.1038/leu.2017.265. Epub 2017 Aug 18. PMID 28819280
- [Background] Schramm F, Zimmermann M, Jorch N, Pekrun A, Borkhardt A, Imschweiler T, Christiansen H, Faber J, Feuchtinger T, Schmid I, Beron G, Horstmann MA, Escherich G. Daunorubicin during delayed intensification decreases the incidence of infectious complications - a randomized comparison in trial CoALL 08-09. Leuk Lymphoma. 2019 Jan;60(1):60-68. doi: 10.1080/10428194.2018.1473575. Epub 2018 Jul 3. PMID 29966458
- [Background] Mondelaers V, Suciu S, De Moerloose B, Ferster A, Mazingue F, Plat G, Yakouben K, Uyttebroeck A, Lutz P, Costa V, Sirvent N, Plouvier E, Munzer M, Poiree M, Minckes O, Millot F, Plantaz D, Maes P, Hoyoux C, Cave H, Rohrlich P, Bertrand Y, Benoit Y; Children-s Leukemia Group (CLG) of the European Organization for Research and Treatment of Cancer (EORTC). Prolonged versus standard native E. coli asparaginase therapy in childhood acute lymphoblastic leukemia and non-Hodgkin lymphoma: final results of the EORTC-CLG randomized phase III trial 58951. Haematologica. 2017 Oct;102(10):1727-1738. doi: 10.3324/haematol.2017.165845. Epub 2017 Jul 27. PMID 28751566
- [Background] Vora A, Goulden N, Wade R, Mitchell C, Hancock J, Hough R, Rowntree C, Richards S. Treatment reduction for children and young adults with low-risk acute lymphoblastic leukaemia defined by minimal residual disease (UKALL 2003): a randomised controlled trial. Lancet Oncol. 2013 Mar;14(3):199-209. doi: 10.1016/S1470-2045(12)70600-9. Epub 2013 Feb 7. PMID 23395119
- [Background] Pieters R, de Groot-Kruseman H, Van der Velden V, Fiocco M, van den Berg H, de Bont E, Egeler RM, Hoogerbrugge P, Kaspers G, Van der Schoot E, De Haas V, Van Dongen J. Successful Therapy Reduction and Intensification for Childhood Acute Lymphoblastic Leukemia Based on Minimal Residual Disease Monitoring: Study ALL10 From the Dutch Childhood Oncology Group. J Clin Oncol. 2016 Aug 1;34(22):2591-601. doi: 10.1200/JCO.2015.64.6364. Epub 2016 Jun 6. PMID 27269950
- [Derived] Toksvang LN, Als-Nielsen B, Bacon C, Bertasiute R, Duarte X, Escherich G, Helgadottir EA, Johannsdottir IR, Jonsson OG, Kozlowski P, Langenskjold C, Lepik K, Niinimaki R, Overgaard UM, Punab M, Raty R, Segers H, van der Sluis I, Smith OP, Strullu M, Vaitkeviciene G, Wik HS, Heyman M, Schmiegelow K. Thiopurine Enhanced ALL Maintenance (TEAM): study protocol for a randomized study to evaluate the improvement in disease-free survival by adding very low dose 6-thioguanine to 6-mercaptopurine/methotrexate-based maintenance therapy in pediatric and adult patients (0-45 years) with newly diagnosed B-cell precursor or T-cell acute lymphoblastic leukemia treated according to the intermediate risk-high group of the ALLTogether1 protocol. BMC Cancer. 2022 May 2;22(1):483. doi: 10.1186/s12885-022-09522-3. PMID 35501736